CLINICAL TRIAL: NCT04612972
Title: Ensayo Clínico de Fase III, Aleatorio, Doble Ciego y Controlado Con Placebo Paralelo, Para Evaluar la Seguridad y la Eficacia Protectora de la Vacuna Inactivada Contra el SARS-CoV-2 en la Población Sana de 18 años o más, en Perú
Brief Title: Efficacy, Safety and Immunogenicity of Inactivated SARS-CoV-2 Vaccines (Vero Cell) to Prevent COVID-19 in Healthy Adult Population In Peru Healthy Adult Population In Peru
Acronym: Covid-Peru
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: National University of San Marcos, Peru (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UPeruanaCH
Record Dates: First submitted 2020-08-18; First posted 2020-11-03 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Arm 1:Investigational vaccine 1:
  Inactivated SARS-CoV-2 vaccine (Vero cell) Manufacturer: Wuhan Institute of Biological Products Co., Ltd. Wuhan Institute of Virology, Chinese Academy of Sciences Specification: 200WU/dose for per human use, 0.5 mL/ dose
  Arm 2: Investigational vaccine 2:
  Inactivated SARS-CoV-2 vaccine (Vero cell) Manufacturer: Beijing Institute of Biological Products Co., Ltd. Specification: 4μg/dose for per human use, 0.5 mL/ dose
  Arm 3: Placebo Product name: Placebo/Aluminum Adjuvant of Inactivated SARS-CoV-2 vaccine Active Ingredient: None; Virus Contents: None Adjuvant: aluminum hydroxide Manufacturer: Wuhan Institute of Biological Products Co., Ltd. Specification: 0.5 mL/ dose, 0.5mL for per human use
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Researchers and participants are masked to Intervention group. Individual syringes are coded with a consecutive number only
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Investigational vaccine 1. Wuhan (Experimental): Inactivated SARS-CoV-2 vaccine (Vero cell); 200WU/dose for per human use, 0.5 mL/ dose; Intramuscular injection; Two doses: one dose/21-28 days; 4000 participants per arm
  Interventions: Biological: Inactivated SARS CoV 2 vaccine (Vero cell) Wuhan/Beijing/Placebo
- Investigational vaccine 2. Beijing (Experimental): Inactivated SARS-CoV-2 vaccine (Vero cell); 4μg/dose for per human use, 0.5 mL/ dose; Intramuscular injection; Two doses: one dose/21-28 days; 4000 participants per arm
  Interventions: Biological: Inactivated SARS CoV 2 vaccine (Vero cell) Wuhan/Beijing/Placebo
- Placebo/Aluminum Adjuvant of Inactivated SARS CoV (Placebo Comparator): Placebo/Aluminum Adjuvant of Inactivated SARS-CoV-2 vaccine; Active Ingredient: None; Virus Contents: None; Adjuvant: aluminum hydroxide; Specification: 0.5 mL/ dose, 0.5mL for per human use; Intramuscular injection; Two doses: one dose/21-28 days; 4000 participants per arm
  Interventions: Biological: Inactivated SARS CoV 2 vaccine (Vero cell) Wuhan/Beijing/Placebo

INTERVENTIONS:
Biological: Inactivated SARS CoV 2 vaccine (Vero cell) Wuhan/Beijing/Placebo — This clinical trial is conducted in randomized, blind, placebo controlled design Total sample size is 12 000, which are randomly allocated into investigational vaccine 1, investigational vaccine 2 and placebo control group.

SUMMARY:
This is a multicenter, randomized, double blind, parallel placebo controlled, phase 3 clinical trial to evaluate the protective efficacy, safety and immunogenicity of inactivated SARS-CoV-2 vaccines in healthy population 18 years old and above.

DETAILED DESCRIPTION:
Product characteristics:

WIBP:

The inactivated SARS CoV 2 Vaccine (Vero cell) is prepared by inoculating Verda Reno cells (Vero cell) with SARS CoV 2 WIV04 strain, culturing, harvesting, inactivating, clarifying, concentrating, second inactivating, purifying and adding aluminum hydroxide adjuvant BIBP: The inactivated SARS CoV 2 Vaccine (Vero cell) is prepared by inoculating Verda Reno cells (Vero cell) with SARS CoV 2 HB02 strain, culturing, harvesting, inactivating, clarifying, concentrating, purifying and adding aluminum hydroxide adjuvant. After vaccination, the body can produce immune response to prevent diseases caused by SARS CoV 2.

Primary objective To evaluate the protective efficacy of inactivated SARS CoV 2 Vaccine (Vero Cell) after full course of immunization in preventing diseases caused by the SARS CoV 2 in healthy subjects aged 18 years old and above.

Study design:

This clinical trial is conducted in randomized, blind, placebo-controlled design. Total sample size is 12,000, which are randomly allocated into investigational vaccine 1, investigational vaccine 2 and placebo control group. Subjects with compatible symptoms, will be excluded.

Immunization schedule: 2-doses of investigational vaccine or placebo are inoculated to the deltoid muscle of the upper arm according to the Day 0 and day 21 (window for both days + 7 days), immunization schedule.

Safety observation After each dose of vaccination, the subject is observed for 30 minutes on site, and local and systemic adverse events are collected. Within 0-30 21/28 days, the local and systemic reactions of the subjects are actively followed up and recorded on the. telephone follow-up contact form. Serious adverse events (SAE) will be daily monitored within 12 months after vaccination, and followed up, recorded and reported as required.

Observation of efficacy After the subjects are enrolled in the group, the monitoring of SARS-CoV-2 infection cases will begin Planned and active follow-up is carried out on the subjects, and a monitoring network is established in local medical and health institutions to monitor SARS-CoV-2 infection-like cases in the subjects. Those diagnosed as suspected cases by clinicians will be studied as epidemiological case, including nasopharyngeal swabs, sputum and/or other lower respiratory secretions, venous blood in acute and convalescent stages are collected. SARS-CoV-2 nucleic acid will be tested by RT-PCR method, and/or viral gene sequencing. Subjects with positive nucleic acid, or/and convalescent serum antibodies increased 4 fold or more than acute phase serum are confirmed cases of COVID-19. (refer to case monitoring operation manual).

The incidence of confirmed SARS-CoV-2 disease in the three groups of study samples is calculated and the epidemiological protection rate and confidence interval of SARS-CoV-2 inactivated vaccines against SARS-CoV-2 disease are analyzed.

Immunogenicity observation:

Immunogenicity (antibody response to inactivated SARS-CoV-2 vaccine / placebo) will be evaluated in subjects V00001-V12000 on 14 days after 2nd dose (day 35) and 360 days after 2nd dose (day 381). Subgroups of 1200 participants will be registered on 28 days after 2nd dose (days 49), 180 days after 2nd dose ( day 201), to better precise the peak of neutralizing antibodies

Case definition:

Cases will be further classified as:

Asymptomatic cases: No symptoms developed for 14 consecutive days after positive PCR testing.

Confirmed cases: On the basis of the clarification of the suspected case, the COVID-19 PCR diagnosis is positive, or IgG antibodies in convalescent sera four times higher than baseline.

Confirmed mild COVID-19 cases: The clinical symptoms were mild, and there was no sign of pneumonia on imaging.

Confirmed moderate COVID-19 cases: Showing fever and respiratory symptoms with radiological findings of pneumonia.

Confirmed severe COVID-19 cases: Confirmed COVID-19 case meeting any one of the following criteria:

* Respiratory distress (RR≥30 breaths/min);
* Oxygen saturation≤93% at rest;
* Arterial partial pressure of oxygen (PaO2)/ fraction of inspired oxygen (FiO2)≦300mmHg (1mmHg=0.133kPa);
* The clinical symptoms progressively worsened, and the chest imaging showed >50% obvious lesion progression within 24-48 hours.

Confirmed Critical COVID-19 cases: Confirmed COVID-19 case meeting any one of the following criteria:

* Respiratory failure and requiring mechanical ventilation;
* Shock;
* With other organ failure that requires ICU care;
* Death

ELIGIBILITY:
Inclusion Criteria:

* Age range: Healthy subjects aged 18 years old and above
* By asking for medical history and physical examination, the investigator judged that the health condition is well
* Female subjects of childbearing age are not nursing or pregnant at the time of enrolment (negative urine pregnancy test), and do not plan to become pregnant within the first 3 months after enrolment . Effective contraceptive measures have been taken within 2 weeks before inclusion and continued for at least three month s after last dose
* During the whole follow up period of the study, be able and willing to complete the whole prescribed study plan.
* With self ability to understand the research procedures, with informed consent, voluntarily sign an informed consent form, and be able to comply with the requirements of the clinical study protocol.

Exclusion Criteria:

* SARS CoV 2 Infection Confirmed Cases, Suspected Cases or Asymptomatic Infection
* SARS CoV 2 Nucleic acid test positive
* Have a history of SARS , MERS infection (self report, on site inquiry
* Fever (axillary temperature > 37.0 ℃), dry cough, fatigue, nasal obstruction, runny nose, pharyngeal pain, myalgia, diarrhea, shortness of breath and dyspnea occurred within 14 days before vaccination
* Axillary body temperature > 37.0 ℃ before vaccination
* Previous severe allergic reactions to vaccination (such as acute allergic reactions, urticaria, dyspnea, angioneurotic edema or abdominal pain) or allergy to known ingredients of inactivated SARS CoV 2 vaccine have occurred.
* Have a history of convulsion, epilepsy, encephalopathy or mental illness or family history
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.
* Severe liver and kidney diseases, uncontrollable hypertension (systolic blood pressure ≥ 140 mmHg, diastolic blood pressure ≥ 90 mmHg), diabetic complications, malignant tumors, various acute diseases or acute attack period of chronic diseases
* Has been diagnosed with congenital or acquired immune deficiency, HIV infection, lymphoma, leukemia or other autoimmune diseases
* Diseases known or suspected include severe respiratory diseases, severe cardiovascular diseases, liver and kidney diseases, and malignant tumors. - Hist ory of coagulation dysfunction (e.g. Coagulation factor deficiency, coagulation disease)
* Receiving anti TB therapy
* Patients receiving immunotherapy or inhibitor therapy within 3 months (continuous oral or infusion for more than 14
* Live attenuated va ccine is inoculated within 1 month before this vaccination , other vaccines are inoculated within 14 days before this vaccination
* Received blood products within 3 months before this vaccination
* Received other research drugs within 6 months before this vacc ination
* Investigator judged other circumstances that are not suitable for this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12000 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Proportion of confirmed Covid-19 cases in the two vaccine groups and the placebo group. | One year beginning on day 14 after the second dose of immunization
  Protective effect against COVID 19, after 14 days following the full course of vaccination among healthy population aged 18 years old and above. Comparison of the proportions of confirmed Covid-19 cases in the two vaccine groups and the placebo group. All confirmed cases are all confirmed by DSMB blind examination.

SECONDARY OUTCOMES:
Proportion of severe cases of SARS CoV 2 pneumonia and deaths in the two vaccine groups and the placebo group. | One year beginning on day 14 after the second dose of immunization
  To evaluate the protective effect after 14 days following 2 doses of immunization of preventing severe cases of SARS CoV 2 pneumonia and deaths caused by COVID 19, among healthy population aged 18 years old and above. Comparison of the proportions of severe cases of SARS CoV 2 pneumonia and deaths in the two vaccine groups and the placebo group.
Incidence of any adverse reactions/events | 12 months
  Observe the incidence of any adverse reactions/events within 30 minutes after each dose of vaccine Observe the incidence of adverse reactions/events at 0 ~ 7 days and 8 ~ 21/30 days after each dose of vaccine. Observe the incidence of serious adverse events (SAE) from the beginning of the first dose to 12 months after the whole course of immunization.

OTHER OUTCOMES:
Comparison of levels of neutralizing antibodies in infected versus non infected participants | After 14 days after 2 doses of immunization
  To explore the protective level of anti-SARS-CoV-2 neutralizing antibody against diseases caused by SARS-CoV-2 infection.
Number of ADE/VED cases | 28days after full course of immunization.
  The occurrence of ADE/VED after immunization.
4-fold growth rate, GMT and GMI of anti-SARS-CoV-2 neutralizing antibody at day 28 | 28days after full course of immunization.
  To evaluate the 4-fold growth rate, GMT and GMI of anti-SARS-CoV-2 neutralizing antibody 28days after full course of immunization.
GMT of anti-SARS-CoV-2 neutralizing antibody at 6 and 12 months | 6th month and 12th month after 2 doses of immunization.
  The GMT of anti-SARS-CoV-2 neutralizing antibody in 6th month and 12th month after 2 doses of immunization.

CONTACTS AND LOCATIONS:
Overall Officials: Coralith Garcia, MD, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (1):
- Av. Honorio Delgado 430, Urb. Ingeniería, San Martín de Porres, Lima region, Peru